CLINICAL TRIAL: NCT01197898
Title: Evaluation of the Edge of Non-Healing Cutaneous Ulcers Following Debridement With Collagenase Santyl Ointment
Brief Title: Wound Edge Changes Following Treatment With Santyl
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 017-101-09-029
Record Dates: First submitted 2010-08-26; First posted 2010-09-09 (Estimated); Results first posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-04

CONDITIONS: Diabetic Foot Ulcers; Diabetic Foot Wounds
Keywords: Diabetic; Foot; Ulcers; Wounds
MeSH Terms: conditions — Diabetic Foot; Ulcer; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagenase Santyl (Experimental): Ointment applied once daily
  Interventions: Biological: Collagenase Santyl Ointment
- Vehicle Base (Placebo Comparator): Applied once daily
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Biological: Collagenase Santyl Ointment — Topical daily application
  Arms: Collagenase Santyl
Other: Placebo Comparator — Topical daily application
  Arms: Vehicle Base

SUMMARY:
The goal of this study is to evaluate changes in the healing tissue of diabetic foot wounds following 14 days of treatment with Santyl or its vehicle base.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, subjects must meet the following inclusion criteria:

* Subjects should be presenting for the first time with a complaint of a non-healing wound, or may have failed one or more prior inadequate therapies. To improve homogeneity in the group studied, subjects with large wounds, complicated wounds, wounds of long duration, or who have failed multiple attempts at healing in which additional known critical variables were addressed (debridement, off loading, wound moisture control, wound infection control, blood glucose control, and/or adequate local blood supply) will be excluded.
* Provide written informed consent.
* Subjects 18 years of age or older, of either sex and of any race, with an existing diagnosis of Type I or Type II Diabetes Mellitus.
* Presenting for the first time with a complaint of a non-healing wound, or may have failed one or more prior inadequate therapies but not including therapies generally reserved for chronic wounds (i.e., debridement, off loading, wound moisture control, wound infection control, blood glucose control, and/or adequate local blood supply).
* Willing to attend all required study visits, and in the opinion of the Investigator, able to properly follow instructions regarding daily dressing changes (dressing changes may be done by a third party, who must agree to perform these daily).
* Body Mass Index less than or equal to 40
* A foot wound which meets the following criteria:

  * Time since initial skin breakdown 56 - 112 days
  * Wagner† Grade 1
  * Area between 0.75 and 3.0 cm2, inclusive
  * Located on plantar surface of midfoot or forefoot, dorsum of foot, or a post-amputation wound
  * Non-infected based on clinical assessment
* Adequate blood supply to the affected foot, defined as meeting a transcutaneous oxygen pressure(TcPO2) measured using standard technique and within 4 cm of the wound of greater than or equal to 35 mmHg.
* Blood chemistry and hematology values as follows, using local lab normal ranges unless otherwise specified:

  * Blood Glycated Hemoglobin (HbA1C) 6.5 - 10.5%
  * Blood Glucose less than or equal to 180 mg/dL
  * Blood Hemoglobin, Hematocrit, Red Blood Cell count within normal limits
  * Serum Sodium, Potassium, Calcium, Phosphorus, Carbon Dioxide (CO2) within normal limits
  * Serum Albumin greater than or equal to 2.0 g/dL, serum Pre-Albumin greater than or equal to 15 mg/dL
  * Alanine Transaminase (ALT), Aspartate Transaminase (AST), Gamma Glutamyl Transpeptidase (GGT) less than or equal to 2.0 x Upper Limit of Normal (ULN)
  * Blood Urea Nitrogen, Total Bilirubin, Creatinine less than or equal to 1.5 x ULN
* Wound is able to be off-loaded, if indicated. † Wagner Grade 1 = Superficial ulcer, partial or full-thickness, but not involving underlying fat, fascia, tendon, muscle or bone.

Exclusion Criteria:

Subjects meeting any of the following criteria during the screening period will be excluded from the study:

* Contraindications or hypersensitivity to the use of the study medications or their components
* Therapy with another investigational agent within thirty (30) days of Visit 1.
* Calluses or maceration of periwound area which would interfere with successful biopsy of the wound edge.
* Undermining or tunneling of the target wound.
* Evidence of osteomyelitis on screening roentgenogram of the target foot.
* Coagulation defect or bleeding disorder which, in the opinion of the Investigator, will make the biopsy procedures too risky.
* The Medical Monitor may declare any subject ineligible for a valid medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Art J Tallis, DPM, Principal Investigator — Associated Foot & Ankle Specialists
Locations (1):
- Associated Foot and Ankle Specialists, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Type I or II diabetes mellitus and a non-healing foot ulcer including postamputation wounds and wounds on the dorsum of the foot.
Groups:
- Collagenase Santyl Ointment: Applied once daily
  Collagenase Santyl Ointment : Topical daily application
- Vehicle Base: Applied once daily
  Placebo Comparator : Topical daily application
Period: Overall Study
Arm/Group | Collagenase Santyl Ointment | Vehicle Base
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collagenase Santyl Ointment | Vehicle Base | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 4 | 4
  >=65 years | 5 | 1 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 72.4 (8.3) | 50.6 (10.2) | 61.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Extent of Presence/Absence of Epithelial Tongue.
Description: The results were found to be inconclusive due to the small number of biopsy specimens of sufficient quality for analysis. Four of the 10 subjects enrolled were not evaluable due to poor biopsy quality.
Time Frame: 28 Days
Population: Goal was to complete 10 subjects in an allocation ratio of 1:1 for Santyl vs. placebo. Since this was an exploratory study, the sample size was arbitrary.
Measure: Number; unit: participants
Arm/Group | Collagenase Santyl Ointment | Vehicle Base
Number analyzed (Participants) | 3 | 3
participants | NA — The results were found to be inconclusive due to the small number of biopsy specimens of sufficient quality for analysis. | NA — The results were found to be inconclusive due to the small number of biopsy specimens of sufficient quality for analysis.

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Collagenase Santyl Ointment | Vehicle Base
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collagenase Santyl Ointment (N=5) | Vehicle Base (N=5)
Acute Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) — SAE judged to be not related to test article by the Investigator

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release.